CLINICAL TRIAL: NCT07265947
Title: A Phase 2A/B, Multi-center, Open-Label Study Evaluating the Efficacy and Safety of Dabogratinib (TYRA-300) in Participants With Low Grade Upper Tract Urothelial Carcinoma (SURF303)
Brief Title: Phase 2A/B Efficacy and Safety of Dabogratinib in Participants With Low Grade Upper Tract Urothelial Carcinoma
Acronym: SURF303
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tyra Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TYR300-203; 2025-523539-20-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-19; First posted 2025-12-05 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Low Grade Upper Tract Urothelial Carcinoma
Keywords: Low-grade UTUC; Upper Tract Urothelial Carcinoma; Low Grade Upper Tract Urothelial Carcinoma; FGFR Gene Amplification; FGFR Gene Alteration; FGFR Gene Alterations; FGFR3 Mutation; FGFR3 Mutations; FGFR3 Gene Fusions

STUDY DESIGN:
Intervention Model Description: Two doses will be explored in Phase 2A (Dose Cohort A (DCA) 80 mg QD) and Dose Cohort B (DCB) 60 mg QD) in parallel design, enrolled by 1:1 randomization. Once the optimized dose is identified, additional participants may be enrolled at the recommended Phase 2B dose to further investigate the efficacy, safety, PK, and therapeutic activity of dabogratinib prior to the official initiation of Phase 2B enrollment. Up to 130 participants may be enrolled in Phase 2A.
  In Phase 2B, approximately 100 participants will be enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Study Drug Dose Cohort A (DCA) 60mg (Experimental): Dabogratinib (TYRA-300) monotherapy in Participants
  Interventions: Drug: Dabogratinib (TYRA-300) 60mg
- Study Drug Dose Cohort B (DCB) 80mg (Experimental): Dabogratinib (TYRA-300) monotherapy in Participants
  Interventions: Drug: Dabogratinib (TYRA-300) 80mg
- Possible Study Drug Dose Cohort C (DCC) TBD mg (Experimental): Dabogratinib (TYRA-300) monotherapy in Participants
  Interventions: Drug: Dabogratinib (TYRA-300) TBD

INTERVENTIONS:
Drug: Dabogratinib (TYRA-300) 60mg — Self-administered 60mg dose Oral tablet(s) given daily
  Other Names: TYRA-300
  Arms: Study Drug Dose Cohort A (DCA) 60mg
Drug: Dabogratinib (TYRA-300) 80mg — Self-administered 80mg dose Oral tablet(s) given daily
  Other Names: TYRA-300
  Arms: Study Drug Dose Cohort B (DCB) 80mg
Drug: Dabogratinib (TYRA-300) TBD — To be determined: Self-administered Oral tablet(s) given daily
  Other Names: TYRA-300
  Arms: Possible Study Drug Dose Cohort C (DCC) TBD mg

SUMMARY:
A Phase 2A/B study of Dabogratinib (TYRA-300) in Low Grade Upper Tract Urothelial Carcinoma

DETAILED DESCRIPTION:
A Phase 2A/B, Multi-center, Open-Label Study Evaluating the Efficacy and Safety of Dabogratinib (TYRA-300) in Participants with Low Grade Upper Tract Urothelial Carcinoma (SURF303)

ELIGIBILITY:
1. Participants ≥ 18 years of age at the time of informed consent and willing and able to comply with all required study procedures
2. Confirmed LOW RISK LG UTUC (both favorable and unfavorable) per AUA
3. At least 5mm of marker lesion left behind
4. Participants must have previous genomic report or archival/fresh tissue in addition to urine sample for retrospective genomic testing
5. Identification of marker lesion(s) within 8 weeks prior to randomization (refer to Inclusion Criterion #2)
6. If synchronous NMIBC, NMIBC must be fully resected and low-grade Ta or T1
7. No prior BCG administration within 1 year of date of consent.
8. No intravesical chemotherapy within 8 weeks prior to C1D1 (including UGN-101).
9. No systemic chemotherapy within 3 months prior to C1D1
10. ECOG 0-2
11. Pathology consists of pure urothelial carcinoma
12. Adequate bone marrow, liver, and renal function:

    1. i. Absolute neutrophil count (ANC) ≥1,500/mm3 ii. Platelet count ≥75,000/mm3 iii. Hemoglobin ≥10.0 g/dL
    2. i. Total bilirubin ≤ ULN ii. Alanine aminotransferase (ALT) ≤ ULN iii. Aspartate aminotransferase (AST) ≤ ULN
    3. Estimated glomerular filtration rate >60 mL/min
    4. Serum Phosphate level ≤ ULN prior to starting treatment
    5. International normalized ratio (INR) ≤1.5 × ULN

Exclusion Criteria:

1. Evidence or any features of high grade (HG) UTUC
2. History of carcinoma in situ (CIS)
3. History of prostatic urethral involvement
4. Current or previous history of muscle invasive bladder cancer
5. Current or previous history of lymph node positive and/or metastatic bladder cancer
6. Evidence of squamous cell carcinoma, adenocarcinoma or undifferentiated carcinoma or small cell of the bladder
7. Currently receiving systemic cancer therapy (cytotoxic or immunotherapy)
8. Current or prior history of pelvic external beam radiotherapy for bladder cancer
9. Current or history of receiving a prior FGFR inhibitor
10. Systemic immunotherapy within 6 months prior to randomization
11. Treatment with an investigational agent within 30 days or 5 half-lives from randomization, whichever is shorter; compounds with an unknown half-life will be default to 30 days.
12. Prior treatment with an intravesical or intracavitary agent within 8 weeks of C1D1.
13. Current evidence of central serous retinopathy or retinal pigmented epithelial detachment of any grade at time of baseline examination.
14. Requiring use of medications that are potential inhibitors or inducers of CYP3A (prohibited list of medications)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of Dabogratinib in LG UTUC FGFR3+ participants (proportion of participants with a CR within 6 months out of all LG UTUC FGFR3+ participants) | within 6 months
  Complete response (CR) rate

SECONDARY OUTCOMES:
To assess the efficacy of Dabogratinib in LG UTUC in all participants (proportion of participants with a CR within 6 months out of all LG UTUC participants) | at 6 months
  Complete Response (CR) rate
Duration of Response (DOR)(median time for CR duration in those participants who achieve a CR) | up to 36 months
Complete Response (proportion of participants who continue to have a CR at 12 and 24 months) | at 12 and 24 months
Safety and tolerability of dabogratinib | Up to 2 years
  Incidence rate and severity of adverse events
Rate of renal preservation after treatment with dabogratinib | Up to 2 years
  Proportion of participants who did not undergo a nephrectomy or nephroureterectomy
Change from unresectable UTUC to resectable UTUC | Up to 2 years
  Proportion of participants with unresectable disease at baseline who convert to resectable disease on dabogratinib, as assessed by the Investigator

CONTACTS AND LOCATIONS:
Overall Officials: Erik T. Goluboff, MD, MBA, Study Chair — Tyra Biosciences, Inc
Locations (1):
- Urology Associates, P C, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No